CLINICAL TRIAL: NCT03618394
Title: Early Bone Turnover Markers in Relation to Parenteral Nutrition Regimens
Brief Title: Bone Turnover and Parenteral Nutrition
Status: Completed | Type: Observational
Sponsor: Iaso Maternity Hospital, Athens, Greece (Other)
Collaborators: Harokopio University (Other); National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Panos Papandreou, Clinical Pharmacist, PharmD, Iaso Maternity Hospital, Athens, Greece
Other Study IDs: 29042015
Record Dates: First submitted 2018-07-25; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Bone Turnover Rate Disorder
Keywords: preterms; parenteral; lipid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoflipid: premature neonates receiving MCT/ω-3-PUFA-containing lipid emulsion
  Interventions: Dietary Supplement: MCT/ω-3-PUFA
- Intralipid: premature neonates receiving Soybean Based lipid emulsion
  Interventions: Dietary Supplement: Soybean Based

INTERVENTIONS:
Dietary Supplement: MCT/ω-3-PUFA — lipid emulsion
  Groups: Smoflipid
Dietary Supplement: Soybean Based — lipid emulsion
  Groups: Intralipid

SUMMARY:
Evaluation of changes in biochemical markers of bone metabolism. Fat profile. Evaluation of the overall body development. Assessment of parenteral nutrition protocols.

DETAILED DESCRIPTION:
Osteopenia is very common in premature infants, particularly in preterm infants born at extremely low birth weight This is probably related to inadequate calcium and phosphorus intake, which is considerably less than the accretion of these minerals during the last trimester of pregnancy In addition, severe morbidity during the neonatal period (e.g. bronchopulmonary dysplasia [BPD]), chronic drug therapy (e.g. diuretics and systemic steroids), the need for total parenteral nutrition and prolonged immobility increase the risk of bone demineralization.

Total parenteral nutrition is associated with osteopenia in preterm infants. Insufficient calcium and phosphate are likely causes; aluminum contamination is another possible contributing factor as this adversely affects bone formation and mineralization.

The DHA+ARA-supplemented formulas supported normal growth and bone mineralization in premature infants who were born at <33 wk gestation. Smof lipid emulsion has a high density of this fatty acids, while Intra lipid does not contain any traces of DHA. Evidence has shown that long-chain polyunsaturated fatty acids (LCPUFA), especially the ω-3 fatty acids such as eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) are beneficial for bone health and turnover.

ELIGIBILITY:
Inclusion Criteria:

* gestational age <32 weeks
* birth weight <1500g (VLBW infants)
* in need of Parenteral Nutrition support

Exclusion Criteria:

* >32 weeks of gestation
* chromosomal or other abnormalities
* parenteral nutrition <80% of calorie/fluid needs
* primary liver disease

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Very Low Birth Weight preterm neonates with gestational age <32 weeks
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
change in plasma calcium and osteocalcin levels | 20 days
  Blood sample at 1st or 2nd (within 48 hours of birth) and 20th day of life

SECONDARY OUTCOMES:
change in plasma DHA, EPA levels | 20 days
  Blood sample at 1st or 2nd (within 48 hours of birth) and 20th day of life
cange in plasma OPG levels | 20 days
  Blood sample at 1st or 2nd (within 48 hours of birth) and 20th day of life

CONTACTS AND LOCATIONS:
Locations (1):
- Panos Papandreou, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided